CLINICAL TRIAL: NCT02178514
Title: Do Infants Fed With BabyNes™ System Grow in Agreement With the World Health Organization (WHO) Reference?
Brief Title: BabyNes Nutrition System Growth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11.20.INF
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Growth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formula Feeding group by BabyNes Nutrition System (Experimental): In this arm, all infants will be fed with BabyNes Nutrition System since enrollment until 12 month of age
  Interventions: Other: Formula fed with BabyNes Nutrition System
- Breastfeeding group (No Intervention): used as reference to compare with formula feeding group

INTERVENTIONS:
Other: Formula fed with BabyNes Nutrition System
  Arms: Formula Feeding group by BabyNes Nutrition System

SUMMARY:
Our main research question is: Do infants fed with BabyNes Nutrition System grow in agreement with the WHO reference?

Our second question is: Do infants fed with BabyNes Nutrition System have a metabolic profile closer to breastfed infants?

In order to answer both questions an observational trial will be carried out for 12 months in order to measure weight and to calculate the weight for age z-scores according to the WHO reference.

A breastfeeding group will be used as reference for the metabolic parameters measured in blood of infants from Chinese background.

The effect of the Babynes formulas will be compared to the metabolic values obtained from this breast-feeding reference group.

DETAILED DESCRIPTION:
Design:

12 months-study, with a breastfeeding group for the comparison of metabolic values obtained from a Chinese Reference population.

Number of subjects:

In total, 120 subjects shall be enrolled. 80 subjects will be assigned in formula fed group and 40 subjects to breast feeding group. 20% dropouts are already considered for the sample size of 120.

Product(s) to be tested:

For formula fed group:

* BabyNes 1 months: 0-1 month of age
* BabyNes 2 months: 1-2 months of age
* BabyNes 3-6 months: 3-6 months of age
* BabyNes 7-12 months: 7-12 months of age

For breast feeding group:

* Nan HA 1 once the mothers are no more breastfed from 4 months until 6 months old.
* Nan HA 2 once the mothers are no more breastfed from 6 months until 1 year old.

Amount, dosage, route of administration, duration of study product:

Subjects are included in the study for duration of upto 1 year old of the infant.

For FF group:

From birth to 4 months, they are exclusively fed with the infant formula dispenser (ad libitum).

From 4 months of age they can start diversification but they maintain the adapted infant formula to the age until 12 months.

For BF group:

Mothers are encouraged to exclusively breast feed the infant up to 6 months old or at least until 4 months old. From 4 months of age, or later than 4 months with no more breastfeeding, they can start Nan HA1 / HA 2 (commercial formula) until the age of 12 months. The amount should be suitable for the age and appetite of the infants.

ELIGIBILITY:
Inclusion Criteria:

Healthy newborns, whose mothers had a normal BMI before pregnancy and no diabetes Healthy newborn infant. Full term infant (≥ 37 weeks gestation and ≤ 42 weeks gestation). Birth weight ≥ 2500 g and ≤ 4500 g. Having obtained his/her signed legal representative's informed consent.

For BF group:

* Exclusively breastfed since birth, the infant's mother agrees to exclusively breast feed her infant until at least to 4th month.
* Baby is 3 months (3 months ± 7 days) at enrollment.

For FF group:

* Infant from birth to 21 days of age at the time of enrollment (the 21st day included).
* The infant's mother has voluntarily elected to exclusively formula feed her infant after enrolment.

Exclusion Criteria:

Congenital illness or malformation that may affect normal growth (especially immunodeficiency).

Newborn whose mother's BMI was abnormal (<18.5 or >23.9) at start of pregnancy. Newborn whose mother has diabetes of type-1 or type-2 or other metabolic disorders.

Newborn whose mother has a chronic infectious disease. Newborn whose parents / caregivers cannot be expected to comply with treatment. Newborn currently participating in another nutritional interventional clinical trial (except for vaccination studies).

Max Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
the change in weight-for-age z-score of the WHO Child Growth Standard | from birth to 4 months of age

SECONDARY OUTCOMES:
the Insulin, C-peptide, IGF-1 leptin and ghrelin level | at 4 and 12 months
length and head circumference measures | birth, 1, 2, 4, 6, 9 12 months of age
Body composition: fat mass, lean mass | 4 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China